CLINICAL TRIAL: NCT00466648
Title: Randomized Controlled Trial Comparing Two Different Methods of Laparoscopy Port Closure
Brief Title: Randomized Controlled Trial Comparing Different Closure Methods for Laparoscopic Port Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Presbyterian Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HV-2007
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Laparoscopic Cosmesis
Keywords: laparoscopy, port site, closure, Dermabond
MeSH Terms: interventions — Tissue Adhesives

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Tissue adhesive

SUMMARY:
This study wishes to compare patient satisfaction and cosmesis of two different closure methods of laparoscopic ports. One method uses tissue adhesive (Dermabond) with a deep sub-cutaneous stitch and a Band-Aid dressing. The comparison method uses a 3.o undyed vicryl transcutaneous stitch, with a Bacitracin and Tegaderm dressing.

ELIGIBILITY:
Inclusion Criteria:

* gynecologic laparoscopy patients

Exclusion Criteria:

* known sensitivity to tissue adhesive, antibiotic ointment

Ages: 16 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2007-03; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Del Priore, Principal Investigator — New York Presbyterian Hospital